CLINICAL TRIAL: NCT06101940
Title: A Multicenter Phenotype-Genotype Analysis of Type 1 Myotonic Dystrophy 1 Patients in China
Brief Title: A Multicenter Phenotype-Genotype Analysis of DM1 Patients in China
Status: Enrolling by invitation | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, Professor, Huashan Hospital
Other Study IDs: KY2020-008
Record Dates: First submitted 2021-08-02; First posted 2023-10-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Myotonic Dystrophy 1
Keywords: Observational
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Magnetic Resonance Imaging; Electrocardiography; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples stored in liquid nitrogen and muscle samples preserved in ultra-low temperature freezers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DM1 patients: Patient cohort
  Interventions: Diagnostic Test: MRI scan; Diagnostic Test: Electrocardiography; Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: MRI scan — Brain MRI scan to evaluate the integrity of the nervous system; lower limb muscle MRI scan to evaluate fat infiltration in skeletal muscles of the lower limb
Diagnostic Test: Electrocardiography — Standard 12-lead electrocardiography or Holter monitoring performed to assess cardiac conduction abnormalities and arrhythmias in patients with DM1.
Diagnostic Test: Pulmonary function test — Comprehensive pulmonary function testing including spirometry to assess respiratory muscle weakness and restrictive lung disease in DM1 patients.

SUMMARY:
Myotonic dystrophy 1 (DM1) is an autosomal, dominantly inherited neuromuscular disorder characterized by skeletal muscle weakness, myotonia, cardiac conduction abnormalities, cataracts, and other abnormalities. This disease results from an expansion of a cytosine-thymine-guanine (CTG) trinucleotide repeat in the 3'-untranslated region of the dystrophia myotonica protein kinase (DMPK) gene on chromosome 19. Currently, there is limited phenotype and genotype data available for DM1 patients with Chinese Han ethnicity. Therefore, this study aims to fill this gap and provide complementary data.

DETAILED DESCRIPTION:
This multicenter, prospective, observational study investigates the diagnosis and progression of Myotonic Dystrophy Type 1 (DM1) in Chinese patients through comprehensive data collection. The research protocol includes clinical assessments (strength evaluations, cognitive testing), diagnostic studies (genetic analysis, electromyography), imaging modalities (MRI, echocardiography, electrocardiography), functional evaluations (pulmonary function tests, posture and movement video analysis), and biological sampling (blood and muscle specimens). This integrated approach enables systematic characterization of DM1 manifestations across multiple organ systems, facilitating better understanding of disease progression patterns and potential biomarker identification in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years
* With enough cognitivie ability to understand the content and sign the informed consent form
* With CTG repeats >50 in DMPK gene, revealed by PCR test

Exclusion Criteria:

* Patients with severe mental illness, or severe anxiety and depression
* With comorbidities such as traumatic brain injury and cranial tumors
* A history of alcoholism, psychotropic substance abuse, etc.
* Patients with severe medical conditions and unstable vital signs that cannot tolerate the tests.
* Female in pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be diagnosed and invited to join this trial in each participating neuromuscular diagnostic centers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 10 Metre Walk Test (10MWT) | Baseline, Year 3, Year 5
  The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function

SECONDARY OUTCOMES:
Changes in ESS scale | Baseline, Year 3, Year 5
  The Epworth Sleepiness Scale (ESS) measures the general level of daytime sleepiness. It is a subjective scale ranging from 0 to 24, asking the respondent to rate their propensity to doze off or fall asleep during eight common daily activities to assess the level of daytime sleepiness. A higher score on the ESS indicates a greater likelihood of daytime dozing.
Changes in FSS scale | Baseline, Year 3, Year 5
  The Fatigue Severity Scale (FSS) is a method for evaluating the impact of fatigue on the participant. The FSS questionnaire contains nine statements that rate the severity of the participant's fatigue symptoms, ranging from 7 to 63. A higher score indicates more severe fatigue symptoms in the participant.
Changes in Video Hand Opening Time (vHOT) | Baseline, Year 1, Year 3, Year 5
  The Video Hand Opening Time (vHOT) is a quantitative assessment tool used to measure the time required for patients with myotonic dystrophy to fully open their hands after making a fist. This test evaluates myotonia severity by recording the duration from the initiation of hand opening to complete finger extension. The measurement is performed using video recording to ensure accurate timing. vHOT serves as an objective biomarker for assessing myotonic symptoms and monitoring disease progression in patients with myotonic dystrophy. A longer vHOT indicates more severe myotonia and greater functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Chongbo Zhao, PhD, Study Director — Huashan Hospital
Locations (22):
- China (22):
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First People's Hospital of Yancheng, Yancheng, Jiangsu
  - The First Affiliated Hospital of Nanchang University）, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Gaoxin Hospital, Xi’an, Shanxi
  - Xi'an People's Hospital, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The General Hospital of Western Theater Command, Chengdu, Sichuan
  - Yunnan Provincial People's Hospital, Kunming, Yunnan
  - Huashan Hospital, Shanghai